CLINICAL TRIAL: NCT06568068
Title: The Effect of Preparatory Education on Parental Stress and Attitudes in Parents of Children Entering Early Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Ayşe Metin, Assist. Prof., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 131
Record Dates: First submitted 2024-08-15; First posted 2024-08-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Adolescent Development
Keywords: Adolescent; Parents; Stress; Parent Attitude; Training
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDUCATION GROUP (Experimental): Procedures to be implemented in the Intervention Group:
  The intervention group that will receive training determined after randomization; In Stage 1 An introductory meeting will be held, ERGEP will be announced and educational materials will be distributed. Pretest applications will be done. In Stage 2 A week consisting of four weeks and eight sessions on the following topics determined within the scope of ERGEP Trainings planned to be held in two sessions will be given once.
  Educational Topics:
  1. Developmental periods (oral, anal,a phallic, latent, genital)
  2. Physical, psychological and social changes experienced in girls and boys during adolescence
  3. Being an adolescent parent and healthy communication
  4. Risky behaviors in life and sexual matters during adolescence In Stage 3 At the end of the training, measurement tools will be applied again. In Stage 4 Measuring tools will be repeated after 21 days.
  Interventions: Behavioral: training
- CONTROL GROUP (No Intervention): Procedures to be applied in the Control Group:
  In this group, where no intervention was made, the pretest, interim follow-up and posttest were the same as the intervention group.
  It will be implemented in weeks. It was aimed to present the program to the control group parents at the end of the study.

INTERVENTIONS:
Behavioral: training — The intervention group that will receive training determined after randomization; In Stage 1 An introductory meeting will be held, ERGEP will be announced and educational materials will be distributed. Pretest applications will be done. In Stage 2 A week consisting of four weeks and eight sessions on the following topics determined within the scope of ERGEP Trainings planned to be held in two sessions will be given once.
  1. Developmental periods (oral, anal, phallic, latent, genital)
  2. Physical, psychological and social changes experienced in girls and boys during adolescence
  3. Being an adolescent parent and healthy communication
  4. Risky behaviors in life and sexual matters during adolescence In Stage 3 At the end of the training, measurement tools will be applied again. In Stage 4 Measuring tools will be repeated after 21 days
  Other Names: EDUCATION
  Arms: EDUCATION GROUP

SUMMARY:
Adolescence is defined as a period in which the individual experiences many physiological and psychological changes. Especially in the early adolescence period, the intense emotional ups and downs created by the transition from childhood to adolescence can also lead to difficulties in managing control mechanisms. This period, which has a very important place in vital transition periods, emerges as a period in which the child must receive comprehensive information from his/her parents about the transition to adolescence. However, this process, which challenges the child, also negatively affects the establishment of healthy communication with parents. Therefore, parents cannot talk to their children about these issues, which are "not considered appropriate by society", especially in traditional societies, due to the difficulties brought by the lack of individual information during this process. It is thought that all this chaos of the period will cause intense stress in parents and negatively affect parental attitudes. In this context, it is predicted that the transition to adolescence education program (ERGEP) prepared for parents will positively affect parental stress and parental attitudes.

DETAILED DESCRIPTION:
Adolescence is defined as a period in which the individual experiences many physiological and psychological changes. Especially in the early adolescence period, the intense emotional ups and downs created by the transition from childhood to adolescence can also lead to difficulties in managing control mechanisms. This period, which has a very important place in vital transition periods, emerges as a period in which the child must receive comprehensive information from his/her parents about the transition to adolescence. However, this process, which challenges the child, also negatively affects the establishment of healthy communication with parents. Therefore, parents cannot talk to their children about these issues, which are "not considered appropriate by society", especially in traditional societies, due to the difficulties brought by the lack of individual information during this process. It is thought that all this chaos of the period will cause intense stress in parents and negatively affect parental attitudes. In this context, it is predicted that the transition to adolescence education program (ERGEP) prepared for parents will positively affect parental stress and parental attitudes. This research, which is closely related to Articles 3 and 5 of the Sustainable Development Goals (SDGs), was planned to directly support parents as primary sources in this regard, considering the harms of early adolescent children getting their questions about the issues they need to know and may be curious about during adolescence from the media, websites or unsafe sources. Although it is thought that ERGEP may have many beneficial outputs, this study aims to understand its effects on parental stress and parental attitudes. The study will be conducted as a quasi-experimental research in a state primary school in the Narman district of Erzurum. In the calculation of the sample size, it was planned to conduct the study with 60 parents, 30 intervention and 30 control, considering the class sizes. The Parent Information Form, the Parental Stress Scale (PSS) and the Parental Attitude Scales (4-12 Years) will be used in the collection of data. The data obtained in the study will be analyzed using the SPSS program. Descriptive statistics such as "number, percentage, arithmetic mean, standard deviation" will be used in the evaluation. In order to verify the differences in demographic characteristics between the groups, the chi-square test will be used for categorical variables and the independent sample t-test for continuous variables. The independent sample t-test will be used for the comparison of scale scores between groups, and the paired sample t-test will be used for the comparison within groups. The results of the study will provide an understanding of the effect of ERGEP applied to parents with children in early adolescence on parental stress and parental attitudes. In the event of positive results of the program, the ground will be prepared for the dissemination of ERGEP and the effect of this program on different phenomena can be tested. This study was planned to determine the effect of the transition to puberty preparation education given to parents with children in early adolescence on parental stress and parental attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Not having received such training before
* Being a parent (mother or father) of a 4, 5, 6 and 7th grade student
* Ability to read and write
* Participation is voluntary

Exclusion Criteria:

* Those who cannot attend the entire training program
* Those who did not complete the pre-test, post-test and follow-up measurements
* Those who did not volunteer to participate in the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Parental Stress | 5 MOUNTH
  Change in Parental Stress Parental Stress Scale (PASS): The scale developed by Özmen and Özmen (2012) examines parents' daily It was designed to measure the stress they experience in their relationships with their children. Consisting of 16 questions in total, the scale used A four-point Likert-type rating (Always = 4, Often = 3, Sometimes = 2, Never = 1). The lowest score that can be obtained from the scale is 16, while the highest score is 64. A high score on the scale indicates parental stress. shows that it is high. The internal consistency coefficient of the scale, Cronbach-Alpha, was reported as .85.
Parental Attitude | 5 MOUNTH
  Parental Attitude is Positive Parental Attitude Scales (4-12 Years): The scale developed by Ogelman and Özyürek (2020) was developed to determine the child-rearing attitudes of parents with children aged 4-12. Two subscales were obtained from this study. One of these subscales consists of items reflecting desired attitudes, the other consists of items reflecting undesirable attitudes. The Desired Parental Attitude Scale consists of 14 items, and the Undesirable Parental Attitude Scale consists of 13 items. The high score obtained from these two scales, which are scored and evaluated separately, is interpreted as the dominant attitude related to that scale. The Cronbach Alpha internal consistency coefficient of the scales was reported as 0.810 for the Desired Parental Attitude Scale and 0.748 for the Undesirable Parental Attitude Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Metin, Study Director — kutuphane@erzurum.edu.tr
Locations (1):
- Ayşe Metin, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No